CLINICAL TRIAL: NCT04341909
Title: Trainee Involvement in ERCP Risk Score
Acronym: TIERS
Status: Completed | Type: Observational
Sponsor: Clinical Hospital Colentina (Other)
Collaborators: Policlinico Gemelli, Rome, Italy (Unknown); Cantacuzino Clinical Hospital, Bucharest, Romania (Unknown); Zadar Hospital, Zadar, Croatia (Unknown); University of Belgrade (Other); UHC Zagreb, Zagreb, Croatia (Other Government); Oxford University Hospitals NHS Trust (Other); University of Colorado, Denver, USA (Unknown); Medical University, Sofia, Bulgaria (Unknown); Universitaire Ziekenhuizen KU Leuven (Other); ISUL Hospital, Sofia, Bulgaria (Unknown)
Responsible Party: Principal Investigator, dr. Theodor Alexandru Voiosu, MD, PhD, Clinical Hospital Colentina
Other Study IDs: TIERS
Record Dates: First submitted 2020-04-08; First posted 2020-04-10 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Bile Duct Diseases; Pancreas Cancer
MeSH Terms: conditions — Bile Duct Diseases; Pancreatic Neoplasms | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Trainee Group: Patients who undergo ERCPs with trainee involvement
  Interventions: Procedure: ERCP
- control group: Patients who undergo ERCPs without any trainee involvement
  Interventions: Procedure: ERCP

INTERVENTIONS:
Procedure: ERCP — endoscopic retrograde cholangiopancreatography

SUMMARY:
The study aims to evaluate factors associated with an increased risk of procedure related adverse events (including tecnical failure) of endoscopic retrograde cholangiopancreatography procedures (ERCP) conducted in a teaching setting, with trainee involvement.

DETAILED DESCRIPTION:
The study aims to evaluate factors associated with an increased risk of procedure related adverse events (including tecnical failure) of endoscopic retrograde cholangiopancreatography procedures (ERCP) conducted in a teaching setting, with trainee involvement.

It has previously shown that ERCP procedures with trainee involvement have no additional risk for the patient, but we aim to evaluate whether a subgroup of high-risk procedures can be identified to allow an improvement of the teaching of ERCP, including identifying some high risk features that might indicate that trainee involvement should not be warranted.

Briefly, the study is observational in nature and aims to gather clinical data about the patient and technical data about the procedure (including the degree of trainee involvement( to assess which (if any) procedures carry a higher risk for the patient in a training setting.

data will be gathered using a standard report form completed by the attending endoscopist at the end of each procedure; the form will then be updated at 30days interval with data about potential adverse events.

Patient identity will be protected throughout the study as per regulations in each institution and country; also all patients will sign an informed consent prior to the endoscopic procedure and study enrollment.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing ERCP in the participating centers
* informed consent signed prior to the procedure

Exclusion Criteria:

* refusal to participate / sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all adult patients undergoing ERCP for any indication (diagnostic / therapeutic) in the participating centers
Sampling Method: Probability Sample
Enrollment: 1283 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
any procedure related adverse outcome | 30 days
  including but not limited to cholangitis, perforation, bleeding, technical failure, pancreatitis

CONTACTS AND LOCATIONS:
Overall Officials: theodor voiosu, MD, PhD, Principal Investigator — Colentina Clinical Hospital, UMF Carol Davila Faculty of Medicine
Locations (1):
- Colentina Clinical Hospital, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Voiosu T, Boskoski I, Voiosu AM, Bengus A, Ladic A, Klarin I, Bove V, Busuioc B, Rimbas M, Rustemovic N, Mateescu B, Jovanovic I, Costamagna G. Impact of trainee involvement on the outcome of ERCP procedures: results of a prospective multicenter observational trial. Endoscopy. 2020 Feb;52(2):115-122. doi: 10.1055/a-1049-0359. Epub 2019 Nov 25. PMID 31766060